CLINICAL TRIAL: NCT00813943
Title: Cilengitide in Subjects With Newly Diagnosed Glioblastoma and Unmethylated MGMT Gene Promoter - a Multicenter, Open-label Phase II Study, Investigating Two Cilengitide Regimens in Combination With Standard Treatment (Temozolomide With Concomitant Radiation Therapy, Followed by Temozolomide Maintenance Therapy). [The CORE Study]
Brief Title: Cilengitide, Temozolomide, and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma and Unmethylated Gene Promoter Status
Acronym: CORE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMD121974-012
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Glioblastoma
Keywords: Newly diagnosed Glioblastoma (WHO Grade IV); Cilengitide; Temozolomide; Radiotherapy
MeSH Terms: conditions — Glioblastoma | interventions — Cilengitide; Temozolomide; Radiotherapy

ARMS (3):
- Cilengitide (2-times weekly) + Temozolomide + Radiotherapy (Experimental)
  Interventions: Drug: Cilengitide (2-times weekly); Drug: Temozolomide; Radiation: Radiotherapy
- Cilengitide (5-times weekly) + Temozolomide + Radiotherapy (Experimental)
  Interventions: Drug: cilengitide (5-times weekly); Drug: Temozolomide; Radiation: Radiotherapy
- Temozolomide + Radiotherapy (Active Comparator)
  Interventions: Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cilengitide (2-times weekly) — Cilengitide 2000 milligram (mg) will be administered intravenously twice weekly over 1 hour infusion from Weeks -1 to 77 or until occurrence of progressive disease, unacceptable toxicity, or withdrawal for any other reason. If considered beneficial in the opinion of the Investigator, continuation of cilengitide treatment will be optional in subjects without disease progression and after Week 77 since start of treatment.
  Arms: Cilengitide (2-times weekly) + Temozolomide + Radiotherapy
Drug: cilengitide (5-times weekly) — Cilengitide 2000 milligram (mg) will be administered intravenously 5-times weekly over 1 hour infusion from Weeks -1 to 77 or until occurrence of progressive disease, unacceptable toxicity, or withdrawal for any other reason. If considered beneficial in the opinion of the Investigator, continuation of cilengitide treatment will be optional in subjects without disease progression and after Week 77 since start of treatment.
  Arms: Cilengitide (5-times weekly) + Temozolomide + Radiotherapy
Drug: Temozolomide — Temozolomide (TMZ) 75 milligram per square meter [mg/m^2] will be administered intravenously once daily from Week 1 to 6. From Week 11 onwards, TMZ will be given as maintenance treatment at a dose of 150-200 mg/m^2 for consecutive 5 days every 4 weeks until Week 34 or until disease progression.
Radiation: Radiotherapy — Radiation therapy (RTX) at a dose of 2 gray (Gy) per fraction will be given once daily, 5 days per week from Week 1 to 6, total dose 60 Gy.

SUMMARY:
CORE is a Phase 2 clinical trial in newly diagnosed glioblastoma in subjects with an unmethylated O6-methylguanine-deoxyribonucleic acid methyltransferase (MGMT) gene promoter in the tumor tissue.

The MGMT gene promoter is a section of deoxyribonucleic acid (DNA) that acts as a controlling element in the expression of MGMT. Methylation of the MGMT gene promoter has been found to appear to be a predictive marker for benefit from temozolomide (TMZ) treatment.

In a safety run-in period in dedicated study centers, the safety and tolerability of Cilengitide given as an intense treatment in combination with the first part of standard therapy will be assessed. Thereafter the trial will investigate the overall survival and progression-free survival in subjects receiving two different regimens of Cilengitide in combination with standard treatment versus standard treatment alone.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed histologically proven supratentorial glioblastoma (World Health Organization [WHO] Grade IV, including glioblastoma subtypes, for example, gliosarcoma). The histological diagnosis has to be obtained from a neurosurgical resection of the tumor or by an open biopsy (stereotactic biopsy is not allowed)
2. Tumor tissue specimens from the glioblastoma surgery or open biopsy (formalin-fixed paraffin-embedded) must be available for MGMT gene promoter status analysis and central pathology review
3. Proven unmethylated MGMT gene promoter status (that is, cut-off ratio less than (<) 2 by means of applied test to determine MGMT gene promoter status)
4. Males or females greater than or equal to (>=) 18 years of age
5. Interval of >= 2 weeks but less than or equal to (=<) 7 weeks after surgery or biopsy before first administration of study treatment
6. Available post-operative gadolinium-enhanced magnetic resonance imaging (Gd-MRI) performed within < 48 hours after surgery
7. Stable or decreasing dose of steroids for >= 5 days prior to randomization
8. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1
9. Has to meet 1 of the following recursive partitioning analysis (RPA) classifications:

   * Class III (Age < 50 years and ECOG PS 0)
   * Class IV (meeting one of the following criteria: a) Age < 50 years and ECOG PS 1 or b) Age >= 50 years, underwent prior partial or total tumor resection, Mini Mental State Examination [MMSE] >= 27)
   * Class V (meeting one of the following criteria: a) Age >= 50 years and underwent prior partial or total tumor resection, MMSE < 27 or b) Age >= 50 years and underwent prior tumor biopsy only)
10. Other protocol defined inclusion criteria could apply

Exclusion Criteria:

1. Prior chemotherapy within the last 5 years
2. Prior RTX of the head (except for low dose RTX for tinea capitis)
3. Receiving concurrent investigational agents or has received an investigational agent within the past 30 days prior to the first dose of cilengitide
4. Prior systemic anti-angiogenic therapy
5. Placement of Gliadel® wafer at surgery
6. Planned surgery for other diseases
7. History of recent peptic ulcer disease (endoscopically proven gastric ulcer, duodenal ulcer, or esophageal ulcer) within 6 months of enrollment
8. History of malignancy. Subjects with curatively treated cervical carcinoma in situ or basal cell carcinoma of the skin, or subjects who have been free of other malignancies for >= 5 years are eligible for this study
9. History of coagulation disorder associated with bleeding or recurrent thrombotic events
10. Clinically manifest myocardial insufficiency (New York Heart Association [NYHA] III, IV) or history of myocardial infarction during the past 6 months; or uncontrolled arterial hypertension
11. Inability to undergo Gd-MRI
12. Concurrent illness, including severe infection (for example, human immunodeficiency virus), which may jeopardize the ability of the subject to receive the procedures outlined in this protocol with reasonable safety
13. Subject is pregnant (positive serum beta human chorionic gonadotropin [b-HCG] test at screening) or is currently breast-feeding, anticipates becoming pregnant/impregnating their partner during the study or within 6 months after study participation, or subject does not agree to follow acceptable methods of birth control, such as hormonal contraception, intra-uterine pessar, condoms or sterilization, to avoid conception during the study and for at least 6 months after receiving the last dose of study treatment
14. Current alcohol dependence or drug abuse
15. Known hypersensitivity to the study treatment
16. Legal incapacity or limited legal capacity
17. Presence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
18. Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such
19. Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2009-03; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andriy Markivskyy, MD, Study Director — Merck KGaA, Darmstadt, Germany; Louis B. Nabors, Prof. Dr., Study Chair — University of Alabama at Birmingham
Locations (2):
- Please Contact U.S. Medical Information Located in, Rockland, Massachusetts, United States
- Please Contact the Merck KGaA Communication Center Located in, Darmstadt, Germany

REFERENCES:
- [Derived] Seliger C, Oppong FB, Lefranc F, Chinot O, Stupp R, Nabors B, Gorlia T, Weller M; EORTC Brain Tumor Group. Association of antidepressant drug use with outcome of patients with glioblastoma. Int J Cancer. 2023 Apr 1;152(7):1348-1359. doi: 10.1002/ijc.34344. Epub 2022 Nov 17. PMID 36346112

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participant (informed consent): Mar 2009/Sep 2011. Clinical data cut-off: 07 Feb 2013, Study completion date: Aug 2013.
Pre-assignment Details: Enrolled: 294 screened for eligibility; 29 excluded (mainly due to non-fulfillment of inclusion or exclusion criteria), 265 participants randomized.
Groups:
- Cilengitide (2-times Weekly) + Temozolomide + Radiotherapy: Cilengitide 2000 milligram (mg) twice weekly over 1 hour intravenous infusion from Weeks -1 to 77, Temozolomide (TMZ) 75 milligram per square meter [mg/m^2] intravenously once daily from Weeks 1 to 6, from Week 11 onward, TMZ was given as maintenance treatment at a dose of 150-200 mg/m^2 for consecutive 5 days every 4 weeks until Week 34 and radiotherapy (RTX) at a dose of 2 Gray (Gy) per fraction once daily, 5 days per week from Weeks 1 to 6 or until occurrence of progressive disease, unacceptable toxicity, or withdrawal for any other reason. Continuation of cilengitide treatment after Week 77 was optional in participants without disease progression, If considered beneficial in the opinion of the Investigator.
- Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy: Cilengitide 2000 mg 5-times weekly over 1 hour intravenous infusion from Weeks -1 to 77, TMZ 75 mg/m^2 intravenously once daily from Weeks 1 to 6, from Week 11 onward, TMZ was given as maintenance treatment at a dose of 150-200 mg/m^2 for consecutive 5 days every 4 weeks until Week 34 and RTX at a dose of 2 Gy per fraction once daily, 5 days per week from Weeks 1 to 6 or until occurrence of progressive disease, unacceptable toxicity, or withdrawal for any other reason. Continuation of cilengitide treatment after Week 77 was optional in participants without disease progression, If considered beneficial in the opinion of the Investigator.
- Temozolomide + Radiotherapy: TMZ 75 mg/m^2 administered intravenously once daily from Weeks 1 to 6, from Week 11 onward, TMZ was given as maintenance treatment at a dose of 150-200 mg/m^2 for consecutive 5 days every 4 weeks until Week 34 and RTX at a dose of 2 Gy per fraction once daily, 5 days per week from Weeks 1 to 6 or until occurrence of progressive disease, unacceptable toxicity, or withdrawal for any other reason.
Period: Overall Study
Arm/Group | Cilengitide (2-times Weekly) + Temozolomide + Radiotherapy | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Started | 88 | 88 | 89
Completed | 83 | 83 | 86
Not Completed | 5 | 5 | 3
Not completed — Ongoing at cut-off date | 5 | 5 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all the participants who were randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cilengitide (2-times Weekly) + Temozolomide + Radiotherapy | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy | Total
Number analyzed (Participants) | 88 | 88 | 89 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (9.63) | 55.2 (10.44) | 54.5 (11.64) | 54.8 (10.57)
Gender [Count of Participants; unit: Participants]
  Female | 38 | 38 | 34 | 110
  Male | 50 | 50 | 55 | 155

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Time
Description: The OS time is defined as the time (in months) from randomization to death or last day known to be alive. Participants without event are censored at the last date known to be alive or at the clinical cut-off date, whatever is earlier.
Time Frame: Time from randomization to death or last day known to be alive, reported between day of first participant randomized, that is, Jun 2009 until cut-off date, (07 Feb 2013)
Population: ITT population included all the participants who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cilengitide (2-times Weekly) + Temozolomide + Radiotherapy | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 88 | 88 | 89
Months | 16.3 [13.2 to 18.1] | 14.5 [12.6 to 16.5] | 13.4 [12.2 to 14.3]
Statistical Analysis 1: Comparison: Cilengitide (2-times Weekly) + Temozolomide + Radiotherapy vs Temozolomide + Radiotherapy; Test type: Superiority or Other; p = 0.0328, Log Rank — P-value is not adjusted for multiple testing; Hazard Ratio (HR) = 0.686, 95% CI 2-sided [0.484 to 0.972]
Statistical Analysis 2: Comparison: Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy vs Temozolomide + Radiotherapy; Test type: Superiority or Other; p = 0.3771, Log Rank — P-value is not adjusted for multiple testing; Hazard Ratio (HR) = 0.858, 95% CI 2-sided [0.612 to 1.204]

2. Secondary Outcome: Progression Free Survival (PFS) Time - Investigator and Independent Read
Description: The PFS time is defined as the duration from randomization to either first observation of progressive disease (PD) or occurrence of death due to any cause. Investigator read is the assessment of all imaging by the treating physician at the local trial site. Independent Read is the assessment of all imaging centrally by an Independent Review Committee (IRC).
Time Frame: Time from randomization to disease progression, death or last tumor assessment, reported between day of first participant randomized, that is, Jun 2009 until cut-off date, (07 Feb 2013)
Population: ITT population included all the participants who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cilengitide (2-times Weekly) + Temozolomide + Radiotherapy | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 88 | 88 | 89
Months
  PFS Time: Independent read | 5.6 [3.6 to 5.9] | 5.9 [4.2 to 7.6] | 4.1 [3.7 to 4.7]
  PFS Time: Investigator read | 6.4 [4.2 to 7.9] | 7.5 [5.9 to 8.2] | 6.0 [4.1 to 7.7]

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The Cmax for cilengitide was calculated by non-compartmental analysis using the computer program WinNonlin, Version 6.2. Cilengitide plasma concentrations were determined after dosing on Day 1 (single dose) and Day 5 (repeated doses) of Week 1.
Time Frame: Days 1 and 5 of Week 1
Population: Only "Cilengitide (5-times) + Temozolomide + Radiotherapy" group was analyzed for this outcome measure as per planned analysis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy
Number analyzed (Participants) | 11
nanogram per milliliter (ng/mL)
  Day 1 (Single dose) | 108527 (27197)
  Day 5 (Repeated doses) | 150873 (97220)

4. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) and Terminal Elimination Half-Life (t1/2)
Description: The Tmax and t1/2 for cilengitide were calculated by non-compartmental analysis using the computer program WinNonlin, Version 6.2. Cilengitide plasma concentrations were determined after dosing on Day 1 (single dose) and Day 5 (repeated doses) of Week 1.
Time Frame: Days 1 and 5 of Week 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy
Number analyzed (Participants) | 11
hours
  Tmax: Day 1 (Single dose) | 0.97 (0.34)
  Tmax: Day 5 (Repeated doses) | 1.17 (0.34)
  t1/2: Day 1 (Single dose) | 2.38 (0.8)
  t1/2: Day 5 (Repeated doses) | 2.44 (0.8)

5. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUC [0-infinity]) and Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC [0-24])
Description: The AUC (0-infinity) and AUC (0-24) for cilengitide were calculated by non-compartmental analysis using the computer program WinNonlin, Version 6.2. Cilengitide plasma concentrations were determined after dosing on Day 1 (single dose) and Day 5 (repeated doses) of Week 1.
Time Frame: Days 1 and 5 of Week 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy
Number analyzed (Participants) | 11
hour*ng/mL
  AUC (0-infinity): Day 1 (Single dose) | 280944 (75720)
  AUC (0-infinity): Day 5 (Repeated Doses) | 335263 (105435)
  AUC (0-24): Day 1 (Single dose) | 269941 (82850)
  AUC (0-24): Day 5 (Repeated doses) | 316137 (110425)

6. Secondary Outcome: Plasma Concentration at Pre-dose (Cpre) and Plasma Concentration at End of Infusion (CT)
Description: The Cpre and CT for cilengitide were calculated by non-compartmental analysis using the computer program WinNonlin, Version 6.2. Cilengitide plasma concentrations were determined after dosing on Day 1 (single dose) and Day 5 (repeated doses) of Week 1.
Time Frame: Days 1 and 5 of Week 1
Population: Only "Cilengitide (5-times) + Temozolomide + Radiotherapy" group was analyzed for this outcome measure as per planned analysis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure. One participant had implausible pre-dose concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy
Number analyzed (Participants) | 11
ng/mL
  Cpre: Day 1 (Single dose) | 6372.7 (21135.95)
  Cpre: Day 5 (Repeated doses) | 286.0 (319.05)
  CT: Day 1 (Single dose) | 108045.5 (27981.04)
  CT: Day 5 (Repeated doses) | 157470.0 (99849.26)

7. Secondary Outcome: Apparent Terminal Rate Constant
Description: The apparent terminal rate constant for cilengitide was calculated by non-compartmental analysis using the computer program WinNonlin, Version 6.2. Cilengitide plasma concentrations were determined after dosing on Day 1 (single dose) and Day 5 (repeated doses) of Week 1.
Time Frame: Days 1 and 5 of Week 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: per hour
Arm/Group | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy
Number analyzed (Participants) | 11
per hour
  Day 1 (Single dose) | 0.32 (0.11)
  Day 5 (Repeated doses) | 0.32 (0.11)

8. Secondary Outcome: Mean Residence Time From Time 0 to Infinity (MRT [0-infinity])
Description: The MRT (0-infinity) for cilengitide was calculated by non-compartmental analysis using the computer program WinNonlin, Version 6.2. Cilengitide plasma concentrations were determined after dosing on Day 1 (single dose) and Day 5 (repeated doses) of Week 1.
Time Frame: Days 1 and 5 of Week 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy
Number analyzed (Participants) | 11
hour
  Day 1 (Single dose) | 2.8 (0.71)
  Day 5 (Repeated doses) | 2.9 (0.97)

9. Secondary Outcome: Plasma Clearance (CL)
Description: The CL for cilengitide was calculated by non-compartmental analysis using the computer program WinNonlin, Version 6.2. Cilengitide plasma concentrations were determined after dosing on Day 1 (single dose) and Day 5 (repeated doses) of Week 1.
Time Frame: Days 1 and 5 of Week 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milliliter per minute
Arm/Group | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy
Number analyzed (Participants) | 11
milliliter per minute
  Day 1 (Single dose) | 125.7 (29.93)
  Day 5 (Repeated doses) | 109.3 (36.61)

10. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz) and Apparent Volume of Distribution at Steady State (Vss)
Description: The Vz (after single dose) and Vss (after repeated doses) for cilengitide were calculated by non-compartmental analysis using the computer program WinNonlin, Version 6.2. Cilengitide plasma concentrations were determined after dosing on Day 1 (single dose) and Day 5 (repeated doses) of Week 1.
Time Frame: Days 1 and 5 of Week 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy
Number analyzed (Participants) | 11
liter
  Vz | 24.7 (6.29)
  Vss | 19.2 (8.54)

11. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs, Treatment-Related AEs, Treatment-Related Serious AEs, AEs Leading to Death, Treatment-Related AEs Leading to Death, AEs of Grade 3 or 4 and Treatment-Related AEs of Grade 3 or 4
Description: An AE is defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship. Treatment-emergent AEs are the events between first dose of study drug and up to 28 days after last dose of study treatment. A Serious AE is an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. Treatment-related AEs are the AEs which are suspected to be reasonably related to the study treatment (cilengitide, or radiotherapy, or temozolomide) as per investigator assessment. The severity of AEs was assessed according to the National Cancer Institute-Common Toxicity Criteria (NCI-CTCAE) (Version 3.0): Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening or disabling. Note: Death (Grade 5) was regarded as an outcome.
Time Frame: Time from first dose up to 28 days after last dose of study treatment, reported between day of first participant randomized, that is, Jun 2009 until cut-off date (07 Feb 2013)
Population: Safety population included all the participants who received any dose of study treatment that is Cilengitide, Temozolomide or Radiotherapy. According to trial design safety data in trial arms (Cilengitide vs Control) were collected based on different visit frequency and different safety surveillance period.
Measure: Number; unit: Participants
Arm/Group | Cilengitide (2-times Weekly) + Temozolomide + Radiotherapy | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 89 | 81 | 85
Participants
  AEs | 88 | 80 | 82
  Serious AEs | 47 | 36 | 30
  Treatment-related AEs | 70 | 64 | 56
  Treatment-related serious AEs | 13 | 4 | 5
  AEs leading to death | 8 | 8 | 5
  Treatment-related AEs leading to death | 2 | 2 | 1
  AEs of Grade 3 or 4 | 57 | 47 | 45
  Treatment-related AEs of Grade 3 or 4 | 25 | 19 | 17

12. Secondary Outcome: Number of Participants With AEs Belonging to Standardized Medical Dictionary for Regulatory Activities (MedDRA) Queries (SMQs) Thromboembolic Events and Hemorrhage With NCI-CTC Toxicity Grade 3 or 4
Description: Thromboembolic events (standardized MedDRA query [SMQ]) Grade 3 or 4 AEs encompassed hemiparesis and cerebrovascular accident, pulmonary embolism, and deep vein thrombosis. Thromboembolic events (SMQ) of any grade and of Grade 3 or 4 were generally more frequent in the Cilengitide + Temozolomide/Radiotherapy group than in the Temozolomide/Radiotherapy group but were still in the expected range of this patient population The severity of AEs was assessed according to the National Cancer Institute-Common Toxicity Criteria (NCI-CTCAE) (version 3.0): Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life threatening or disabling. Note: Death (Grade 5) was regarded as an outcome.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Cilengitide (2-times Weekly) + Temozolomide + Radiotherapy | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 89 | 81 | 85
Participants
  SMQ: Thromboembolic events | 17 | 10 | 12
  SMQ:Hemorrhage | 3 | 0 | 1

13. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) and Lab Parameters
Time Frame: as for outcome 11
Population: Any clinically significant abnormal ECG and lab finding was planned to be reported as AE only so they have been captured in the below mentioned adverse event section
Arm/Group | Cilengitide (2-times Weekly) + Temozolomide + Radiotherapy | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Time from first dose up to 28 days after last dose of study treatment, reported between day of first participant randomized, that is, Jun 2009 until cut-off date (07 Feb 2013)
Description: Safety population included all participants who received any dose of study treatment that is Cilengitide, Temozolomide or Radiotherapy. 1 participant who was randomized to cilengitide 5-times weekly, but who actually received Cilengitide 2-times weekly was allocated to the cilengitide 2-times weekly treatment group for the safety population
Arm/Group | Cilengitide (2-times Weekly) + Temozolomide + Radiotherapy | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy | Temozolomide + Radiotherapy
Serious Adverse Events (participants affected / at risk) | 47/89 | 36/81 | 30/85
Other Adverse Events (participants affected / at risk) | 83/89 | 79/81 | 76/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cilengitide (2-times Weekly) + Temozolomide + Radiotherapy (N=89) | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy (N=81) | Temozolomide + Radiotherapy (N=85)
CONVULSION (Nervous system disorders) | 5 | 7 | 3
HEMIPARESIS (Nervous system disorders) | 4 | 3 | 5
EPILEPSY (Nervous system disorders) | 4 | 2 | 1
HEADACHE (Nervous system disorders) | 1 | 1 | 3
BRAIN OEDEMA (Nervous system disorders) | 1 | 0 | 2
CEREBRAL CYST (Nervous system disorders) | 0 | 3 | 0
NEUROLOGICAL DECOMPENSATION (Nervous system disorders) | 0 | 3 | 0
APHASIA (Nervous system disorders) | 0 | 2 | 0
PARTIAL SEIZURES (Nervous system disorders) | 1 | 1 | 0
SOMNOLENCE (Nervous system disorders) | 2 | 0 | 0
CEREBRAL VENTRICLE DILATATION (Nervous system disorders) | 0 | 1 | 0
COGNITIVE DISORDER (Nervous system disorders) | 0 | 1 | 0
DYSARTHRIA (Nervous system disorders) | 1 | 0 | 0
DYSKINESIA (Nervous system disorders) | 0 | 0 | 1
GRAND MAL CONVULSION (Nervous system disorders) | 0 | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 | 0 | 0
HEMIANOPIA (Nervous system disorders) | 1 | 0 | 0
HYDROCEPHALUS (Nervous system disorders) | 0 | 0 | 1
MOTOR DYSFUNCTION (Nervous system disorders) | 0 | 0 | 1
PYRAMIDAL TRACT SYNDROME (Nervous system disorders) | 0 | 1 | 0
RADICULAR PAIN (Nervous system disorders) | 1 | 0 | 0
UNRESPONSIVE TO STIMULI (Nervous system disorders) | 0 | 1 | 0
DISEASE PROGRESSION (General disorders) | 2 | 2 | 0
PYREXIA (General disorders) | 1 | 0 | 3
FATIGUE (General disorders) | 1 | 0 | 2
ASTHENIA (General disorders) | 0 | 1 | 1
CONDITION AGGRAVATED (General disorders) | 1 | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 | 0 | 0
CHEST DISCOMFORT (General disorders) | 0 | 0 | 1
DEVICE MALFUNCTION (General disorders) | 1 | 0 | 0
GAIT DISTURBANCE (General disorders) | 0 | 0 | 1
GENERALISED OEDEMA (General disorders) | 1 | 0 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0 | 0
TERMINAL STATE (General disorders) | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
MEDIASTINAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 4 | 1 | 3
VENOUS THROMBOSIS (Vascular disorders) | 1 | 1 | 0
HYPOTENSION (Vascular disorders) | 1 | 0 | 0
HAEMATOMA (Vascular disorders) | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 1 | 0 | 0
THROMBOSIS (Vascular disorders) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 2 | 0 | 2
BRONCHITIS (Infections and infestations) | 1 | 1 | 0
BACTERIAL SEPSIS (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 1 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0 | 0
MENINGITIS (Infections and infestations) | 1 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 0
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 1 | 0 | 0
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 1 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
NEOPLASM RECURRENCE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
BRAIN NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
BRAIN STEM GLIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
HEAVY CHAIN DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 1 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 1
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 1 | 0
VOMITING (Gastrointestinal disorders) | 2 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1 | 0
FOOD POISONING (Gastrointestinal disorders) | 0 | 1 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 | 0 | 0
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0
PLATELET COUNT DECREASED (Investigations) | 0 | 1 | 2
LIPASE INCREASED (Investigations) | 1 | 0 | 0
AMYLASE INCREASED (Investigations) | 1 | 0 | 0
FIBRIN D DIMER INCREASED (Investigations) | 0 | 0 | 1
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1
BRADYCARDIA (Cardiac disorders) | 1 | 0 | 0
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1 | 0
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 1 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 1 | 1
INSOMNIA (Psychiatric disorders) | 0 | 0 | 1
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 | 0 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0 | 0
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 | 0 | 0
OLIGURIA (Renal and urinary disorders) | 1 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0 | 0
RETINAL ARTERY EMBOLISM (Eye disorders) | 1 | 0 | 0
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SOCIAL STAY HOSPITALISATION (Social circumstances) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cilengitide (2-times Weekly) + Temozolomide + Radiotherapy (N=89) | Cilengitide (5-times Weekly) + Temozolomide + Radiotherapy (N=81) | Temozolomide + Radiotherapy (N=85)
FATIGUE (General disorders) | 27 | 21 | 19
ASTHENIA (General disorders) | 22 | 24 | 11
PYREXIA (General disorders) | 16 | 14 | 8
OEDEMA PERIPHERAL (General disorders) | 9 | 5 | 8
GAIT DISTURBANCE (General disorders) | 3 | 7 | 10
NAUSEA (Gastrointestinal disorders) | 32 | 30 | 30
CONSTIPATION (Gastrointestinal disorders) | 26 | 27 | 27
VOMITING (Gastrointestinal disorders) | 17 | 18 | 21
DIARRHOEA (Gastrointestinal disorders) | 8 | 6 | 2
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 | 5 | 1
STOMATITIS (Gastrointestinal disorders) | 5 | 1 | 2
HEADACHE (Nervous system disorders) | 38 | 32 | 25
CONVULSION (Nervous system disorders) | 8 | 7 | 9
MEMORY IMPAIRMENT (Nervous system disorders) | 7 | 8 | 7
DIZZINESS (Nervous system disorders) | 6 | 5 | 5
APHASIA (Nervous system disorders) | 7 | 3 | 6
TREMOR (Nervous system disorders) | 6 | 5 | 3
DYSGEUSIA (Nervous system disorders) | 6 | 4 | 2
PARAESTHESIA (Nervous system disorders) | 2 | 6 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 9 | 14 | 17
NEUTROPENIA (Blood and lymphatic system disorders) | 11 | 9 | 8
LYMPHOPENIA (Blood and lymphatic system disorders) | 9 | 7 | 7
LEUKOPENIA (Blood and lymphatic system disorders) | 5 | 6 | 7
ANAEMIA (Blood and lymphatic system disorders) | 5 | 9 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 14 | 18 | 11
PRURITUS (Skin and subcutaneous tissue disorders) | 9 | 11 | 5
RASH (Skin and subcutaneous tissue disorders) | 11 | 8 | 3
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4 | 5 | 3
URTICARIA (Skin and subcutaneous tissue disorders) | 2 | 7 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 9 | 19 | 4
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 9 | 3 | 6
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 7 | 3 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 5 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 | 3 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 6 | 2 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 5 | 1
INSOMNIA (Psychiatric disorders) | 12 | 15 | 11
DEPRESSION (Psychiatric disorders) | 12 | 9 | 2
ANXIETY (Psychiatric disorders) | 6 | 7 | 6
URINARY TRACT INFECTION (Infections and infestations) | 6 | 10 | 6
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 | 10 | 5
ORAL CANDIDIASIS (Infections and infestations) | 6 | 6 | 3
NASOPHARYNGITIS (Infections and infestations) | 9 | 5 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 20 | 18 | 18
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 6 | 5 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 | 7 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 3
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 11 | 3 | 3
FALL (Injury, poisoning and procedural complications) | 2 | 5 | 2
HYPERTENSION (Vascular disorders) | 5 | 6 | 3
URINARY INCONTINENCE (Renal and urinary disorders) | 2 | 5 | 3
VISION BLURRED (Eye disorders) | 6 | 2 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All manuscripts and materials relating to Study shall be submitted to Sponsor at least 60 days prior to submitting/presenting and allow Sponsor 60 days for review. If Sponsor requests, any confidential information shall be removed. In multi-center study, any publication shall not be made before the first multi-center publication; provided, however, that if no multi-center publication is made within 1 year from database lock, then Site may publish individually in accordance with this provision.